CLINICAL TRIAL: NCT04660955
Title: Imaging Post-traumatic Osteoarthritis 10-years After ACL Reconstruction
Brief Title: MOON Onsite MRI 10 Years After ACL Reconstruction
Acronym: MRI
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Vanderbilt University Medical Center (Other); Ohio State University (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Xiaojuan Li, Lead Principal Investigator, The Cleveland Clinic
Other Study IDs: 19-573; R01AR075422 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-12-09 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who had ACL reconstruction
  Interventions: Other: No Intervention - Observational study with MRI
- Controls: Controls who have no previous knee injury or surgery, no diagnosis of osteoarthritis
  Interventions: Other: No Intervention - Observational study with MRI

INTERVENTIONS:
Other: No Intervention - Observational study with MRI — 90 minute MRI of the knees

SUMMARY:
In this study, a total of 219 subjects from the MOON nested cohort will be studied at CCF, Vanderbilt and OSU, Table 1. Among them, some will have added MRI during their 10-year visit for the MOON study. Some subjects who finished their 10-year visit for the MOON Onsite study already will be called back to have MRI. PROMs and other information of these subjects will be collected through the MOON study.

DETAILED DESCRIPTION:
In this study, a total of 219 subjects from the MOON nested cohort will be studied at CCF, Vanderbilt and OSU, Table 1. Among them, some will have added MRI during their 10-year visit for the MOON study. Some subjects who finished their 10-year visit for the MOON Onsite study already will be called back to have MRI. PROMs and other information of these subjects will be collected through the MOON study.

In addition, 30 age-, sex- and BMI-matched control subjects (10 from each site) will be recruited and scanned for MRI. PROMs (KOOS, IKDC, Marx, SF-36) will be collected from these controls.

Among the 10 controls recruited locally at CCF, five will also travel to OSU and Vanderbilt to be scanned at the other two sites for cross-validation among the three sites. There will be a separate consent for the 5 controls that will be traveling to each of the 3 sites for the scans. The remaining 25 controls will be tested at only their local site.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in MOON Onsite Study
* 12-33 years old at baseline (22-45 years for this study);
* ACL tear during a sport; no previous knee injury;
* No graft rupture during follow-up;
* No history of surgery on the contralateral knee;
* No MRI contraindications

Exclusion Criteria:

* History of surgery on contralateral knee
* Afraid of enclosed spaces

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This patient cohort include patients who had ACL reconstruction 10 years ago and were recruited in the previous MOON onsite study based on the inclusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Cartilage health status | At 10-years after ACL reconstruction
  Quantitative MRI will be used to quantify cartilage health. Specifically, cartilage MR T1rho and T2 relaxation times will be quantified for cartilage of the knee that had ACL reconstruction, and compared to the contralateral uninjured knee.

SECONDARY OUTCOMES:
Patient reported outcomes | At 10-years after ACL reconstruction
  Pain score (0-100) evaluated using Knee injury and Osteoarthritis Outcome Score (KOOS)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Li, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided